CLINICAL TRIAL: NCT03906981
Title: Dental Plaque Microbiota in Caries-free and Caries-active Arab Children
Brief Title: Dental Plaque Microbiota in Caries-free and Caries-active Children
Status: Completed | Type: Observational
Sponsor: Kuwait University (Other)
Responsible Party: Principal Investigator, Muawia A. Qudeimat, Associate Professor, Kuwait University
Other Study IDs: DD01/14
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Caries; Plaque
MeSH Terms: conditions — Plaque, Amyloid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plaque sample from each subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caries free: 6-9 year old caries free children
  Interventions: Other: Plaque from each subject will be collected but there will be no intervention
- Caries active: 6-9 year-old caries active (>5 dmft/DMFT) children
  Interventions: Other: Plaque from each subject will be collected but there will be no intervention

INTERVENTIONS:
Other: Plaque from each subject will be collected but there will be no intervention — No intervention

SUMMARY:
Dental caries is a polymicrobial infection originally thought to be caused by Streptococcus mutans and Lactobacilli. However, unprecedented developments in modern molecular techniques have demonstrated that several microbial species are associated with the disease in addition to streptococci and lactobacilli. Dental caries initiation and progression is a dynamic process in which demineralization of the tooth structure, as a result of acid production from acidogenic bacteria (due to carbohydrate metabolism) is being counteracted by the remineralization of the tooth surface by strong alkali production by certain bacteria in the dental biofilm. The aim of the present study is to identify the different microbiota in the oral biofilm using new laboratory techniques as well as the levels of salivary proteins in caries-free compared with caries active Arab children.

DETAILED DESCRIPTION:
The objective of this study will be to investigate the dental plaque's microbial diversity using Human Oral Microbe Identification using Next Generation Sequencing (HOMINGS) technology in the mixed dentition as well as the levels of salivary proteins in caries-free compared with caries active Arab children. The study protocol was approved by the Health Science Center Ethical Committee at Kuwait University.

One hundred 6-9 year-old children with caries active and caries-free status will be recruited from randomly selected public schools in Kuwait. After DNA purification from supragingival plaque samples, HOMINGS will be performed. To get an insight into the host factors involved in this complex interplay between the host and the bacteria, stimulated saliva from the study subjects will be analyzed by proteomics. For children in both groups supragingival plaque samples will be collected from the buccal and lingual surfaces of all teeth. After preparing the samples, the aliquots of purified DNA samples will be shipped to The Forsyth Institute for Human Oral Microbe Identification using Next Generation Sequencing (HOMINGS) protocol.

ELIGIBILITY:
Inclusion Criteria:

* Arab 6-9 year old children
* Healthy
* Caries free, dmft/DMFT=0
* Caries Active: dmft/DMFT>5

Exclusion Criteria:

* Children with a systemic disease or any drug use that could affect the microflora of the oral cavity or the salivary gland functions
* History of salivary gland diseases
* Those who received antibiotic therapy during the last 3 months
* Children with severe localized or generalized periodontitis.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pupils from randomly selected public schools
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Dental plaque microbiota profile | 2 months
  Identification of dental plaque microbiota profile using HOMINGS

CONTACTS AND LOCATIONS:
Overall Officials: Muawia A Qudeimat, MDentSci, Principal Investigator — Kuwait University

IPD SHARING:
Plan to Share IPD: Undecided